CLINICAL TRIAL: NCT05946980
Title: hands4health: Hand Hygiene, Water Quality and Sanitation in Primary Health Care Not Connected to Functional Water Supply System: a Cluster-randomized Controlled Trial in Mali and Burkina Faso
Brief Title: hands4health: A Multi-component Intervention on Hand Hygiene in Primary Health Care Facilities in Burkina Faso and Mali
Acronym: h4h
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Terre des Hommes (Unknown); University of Applied Sciences and Arts Northwestern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7F-l 0345.03.01
Record Dates: First submitted 2023-06-16; First posted 2023-07-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hand Hygiene Behavior; Hand Hygiene Effectiveness
Keywords: Hand Hygiene; Behavior Change; Primary Health Care; Primary Schools; Humanitarian Emergency

STUDY DESIGN:
Intervention Model Description: Cluster randomized multi-center controlled trial In each country there is an intervention and control group. The control group will not receive anything until the end of data collection. Afterwards they will receive the intervention as well, improved if needed.
Masking Description: Lab technicians will be masked for hand-rinse sample processing and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm for primary health care facilities in Mali and Burkina Faso (Experimental): This arm receives the multi-component intervention for primary health care facilities described under interventions
  Interventions: Other: Multi-component hand hygiene intervention in primary health care facilities
- Control arm for primary health care facilities in Mali and Burkina Faso (No Intervention): No intervention until the end of the cRCT. After completion of data collection, this arm will receive the same intervention as the intervention arm has received previously.

INTERVENTIONS:
Other: Multi-component hand hygiene intervention in primary health care facilities — Intervention facilities will receive (1), two novel Gravit'eau (https://www.graviteau.ch/) handwashing systems which are locally produced. These systems recycle water for handwashing with gravity through a membrane filter without electricity up to a month. Facilities also receive (2), a behavior change intervention lead by RANAS (https://www.ranasmosler.com/ranas), expert psychologist for behavior change in WASH. They will also receive (3), support to implement WASH FIT (https://washfit.org/#/) in their facilities, a tool developed by WHO to sustainably maintain and improve WASH infrastructure in health care facilities. Additionally, we are recruiting a "circuit rider" responsible for the regular inspection and maintenance of WASH infrastructure. (4), the facilities will receive support for regular water chlorination.
  Other Names: Gravit'eau handwashing system; RANAS behavior change; WASH FIT; Chlorination support
  Arms: Intervention arm for primary health care facilities in Mali and Burkina Faso

SUMMARY:
The goal of this cluster randomized controlled trial is to assess the effectiveness of the hands4health multi-component hand hygiene intervention in patients and health care providers in primary health care facilities in Burkina Faso and Mali. The main question it aims to answer is:

* Can the hands4health multi-component hand hygiene intervention have a positive effect on the health determinants of our study population? Participants will be structurally observed for assessing their handwashing behavior, answer to a self-reported RANAS survey and provide a hand-rinse sample at base line, follow-up and end line. In addition specific pre-defined health outcomes and absenteeism will be tracked with a journal approach in the facilities. Intervention facilities will receive a Gravit'eau handwashing system, a RANAS behaviour change intervention, WASH FIT support, and chlorination support. Control facilities will receive nothing at the beginning, but once all of the data is collected, they will receive the same intervention as the intervention facilities have received. Researchers will compare the intervention and control groups to see if the hands4health intervention has any positive effects on the populations health determinants (e.g. handwashing behavior, perceptions towards hand hygiene, perceived risks, etc.).

DETAILED DESCRIPTION:
The overall project will follow an multi-center cluster-randomized controlled trial (cRCT) design. Prior to this study, the Facility and Evaluation Tool for WASH in Institutions (FACET) has been used to assess the WASH infrastructure of the primary health care facilities (PHCFs) in the study regions. From these PHCFs a subsample was identified which fulfils certain inclusion criteria (see Eligibility).

This subsample was handed over to the local Terre des hommes (Tdh) collaborators who carefully assessed the security situation around the facilities. The Tdh collaborators then chose 24 facilities which are most probable to still be accessible for data collection within the next year. These 24 PHCFs will then be distributed into two arms (intervention vs. control) with stratified randomization using computer-generated randomization code provided by an statistician not involved in any field activities. The intervention arm will receive the full intervention package (see multi-component intervention in health care facilities). The control arm will receive nothing for the duration of the intervention (9 months). Afterwards they will receive the same intervention package with potential improvements identified in the former intervention group.

In the chosen PHCFs all health care workers (HCWs) present at the day of data collection who fulfil the inclusion criteria will be asked to participate in the study. We aim to have as many of the HCWs in all of the Modules 1 and 3 as possible. For Module 2, only a maximum of 10 HCWs per facility will be observed.

The following modules will be used in the cRCT and the overall project to assess the effectiveness of the h4h multi-component intervention: (i) Module 1: Combined RANAS and KAP survey, (ii) Module 2: Structured handwashing observations, (iii) Module 3: Microbiological analysis of hand rinse samples, (iv) Module 4: Diary approach for pre-defined health outcomes, (v) Module 5: Focus Group Discussions (FGDs) and (vi) Module 6: Key informant interviews (KIIs).

The Swiss TPH assessed the health care worker's understanding of hygiene and expected positive and negative impacts of the intervention with Gravit'eau with focus group discussions (FGDs) in 18 facilities in Mali and 9 facilities in Burkina Faso (more facilities are still being investigated). Local collaborators from Tdh and the regional ministries of health were involved from the study's kick-off meeting onwards and are regularly being consulted in bi-weekly meetings and additional ToC workshops led by Skat Foundation. The data collection methods for each module will be described in further detail:

Module 1: Combined RANAS and KAP survey: The survey will be developed through the RANAS approach and will not only include attitude and belief questions, but also target the underlying psychological factors postulated by the RANAS model that are important precursors for effective behaviour change. If needed, this survey will be enriched with additional questions to assess knowledge and self-reported handwashing practices of the participants. The survey will be administered to HCWs three times in total; as a baseline survey before the intervention package, about two months after the intervention and about a year after the baseline survey with the software Open Data Kit (ODK) Central (version 2022.3.1) on Android tablets.

Module 2: Structured handwashing observations: Structured handwashing observations are perceived as a gold standard method to assess handwashing behaviour. Data from Module 1 and the observations can later be combined through a unique ID of the study participants. The observations will be administered with HCWs three times at the same time points as the survey in Module 1.

A trained observer from a Tdh team or the local ministry of health, who normally works in the health care facilities with a different function will visit the facility under the pretence of their usual function. They will be equipped with an observation tool and will follow a healthcare worker for a minimum of one hour at the peak time per PHCF unit for patient visits. The observer will not declare that he/she is observing handwashing practices. Consent will be obtained at a health care facility level, from the director of the health care facility. To avoid making patients feel uncomfortable during sensitive procedures, such as giving birth, only patient visits containing physical examination, injection, and blood sampling will be observed and the patients will be asked for their oral consent prior to entering a room with them.

Module 3: Microbiological analysis of hand rinse samples: Hand rinse samples of HCWs will be collected after the survey with a modified glove juice method as described by Pickering et al. 2010. For the hand rinse sample collection, the participant's hand will be inserted into a 69-oz Whirl-Pak bag (NASCO Corp., Fort Atkinson, WI) filled with 350 mL of clean water. Then, the participant has to shake her/his hand in the water and rub her/his thumb and fingers together for 15 seconds. Afterwards, the data collector will massage the participant's hand through the bag for another 15 seconds. The participant will be provided with a paper towel to dry the hand, once it is retrieved from the bag. Afterwards, the procedure will be repeated with the other hand.

The Whirl-Pak bags containing the samples will be kept on ice in an isolation box and processed within 4 hours of sampling. Membrane filtration will be used to detect colony-forming units (CFUs) of E.Coli and total coliforms. In a field laboratory, the content of the bags will be passed through a 47-mm-diameter 0.45 µm cellulose filter. The filter paper will then be placed on growth media and incubated at 35°C ± 0.5°C for a duration of 24 hours for E.Coli and total coliforms (45). We plan to filter 100 mL per bag to detect CFUs of E.Coli and total coliforms. The exact amount of mL will be established during piloting as the volume used is dependent on the degree of bacterial contamination on the hands. Compact dry plates will be used for the detection of E.coli and total coliforms.

The lower detection limit of CFUs will be calculated by dividing 1 CFU/plate by the filtrate volume and then multiplying it with the total Whirl-Pak volume of 350 mL. The upper detection limit will be calculated by dividing 500 CFUs/plate by the filtrate volume and then multiplying it with the Whirl-Pak volume. For the statistical analysis, the CFUs per hand will be normalized and and log10 transformed.

Module 4: Diary approach for pre-defined health outcomes: Longitudinal data on hygiene-related health outcomes of patients and disease-related absences of HCWs will be collected during 9 months after the intervention in both of the study arms from the cluster-randomized controlled trial with a diary approach. Every time a pre-defined health outcome takes place at facility level, this outcome will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). No patient names or birth dates will be recorded to keep this data fully anonymous. For each health outcome the director will report when it happened, if applicable how long it took, if applicable the number of days of treatment, if known the reason for the outcome and if it was an infection the outcome (recovered, death, unknown). These health outcomes either occur directly at the health care facility, if the facility offers inpatient care, or are reported if the patients report their outcome after a visit (e.g. by calling or re-visiting the facility). The diary consists of one table per month containing all of the different health outcomes and subcategories. Consequently, the HCWs can keep track of these outcomes with a minimal administrative effort. The local study team is still discussing if a paper table, which will be collected once a month will be used, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.

Module 5: Focus Group Discussions: The FGDs will be used to capture the common norms and beliefs of the HCWs. This tool offers many insights in shorter time compared to other qualitative methods such as participatory observation. Data will be collected by a small local team with experience in qualitative data collection and if the security situation allows, by the Swiss TPH PhD student in autumn 2023. The team containing at least one moderator and one observer/note taker will be trained by the PhD student prior to data collection. A field research journal will be used throughout the study to take structured notes and observations of the FGDs. The discussions will be audio recorded and then transcribed into the local language and translated to French or English for further analysis.

Field notes, observation notes and focus group transcripts will be analysed using the framework method with the software MaxQDA (VERBI Software, Marburg, Germany) or NVivo (QSR International, Melbourne, Australia).

Module 6: Key informant interviews: The KIIs will engage with other stakeholders outside of the health care facilities who have an influence on the intervention areas of the project. Some of these key informants will have been identified through the Theory of Change analysis, while others will be suggested by local partners. Individual interviewees were chosen as a tool to gain the insights of these stakeholders, such as people from the ministry of health or the mayor, so that their status does not influence other participant's freedom of speech. The KIIs can be additionally used to inquire further about questions or topics which came up during the FGDs. Further, the format of interviewing can also be used on the health care facility level, in case not enough participants are available for a FGD. The KIIs will take place in autumn 2023.

Interviewers will receive the same training as for the Focus Group Discussions. The interviews will be audio recorded and then transcribed into the local language and translated to French or English for further analysis. In some instances, interviews may be carried out remotely (online) from Switzerland, in French, if it is appropriate. They will be audio recorded, transcribed, and translated if necessary for further analysis.

As the FGD transcripts, the interviews will be analysed using the framework method with the software MaxQDA (VERBI Software, Marburg, Germany) or NVivo (QSR International, Melbourne, Australia).

ELIGIBILITY:
Inclusion Criteria in health care facilities:

Study participants will be health care workers of the primary health care facilities (PHCFs) which were chosen to be included in this study. PHCFs were chosen based on accessibility for the study teams, not having a water source directly connected to the building of the facility, having a maternity ward, having at least five employees and being impacted by conflict. All of the HCWs who are present in the PHCFs of the day of data collection will be invited to participate in the project for Modules 1 and 3.

Inclusion criteria Modules 1-3: HCWs must fulfil all the inclusion criteria:

* Minimum age of 18 years
* HCWs, men and women, who are in direct (body) contact with the patients

During the handwashing observations, HCWs will consult with patients. In order to protect patients, they must meet these inclusion criteria for an observer to be allowed into the consultation room with them:

* Minimum age of 18 years or be accompanied by a legal guardian 18 years or older.
* Going to the SSE for a physical examination, injections/vaccinations or blood test.
* Oral consent to enter the room with them

Inclusion criteria Module 4: As the data will be collected on the health care facility level, all facilities in the project will be included.

Inclusion criteria Module 5:

* HCWs of the intervention facilities
* Minimum age of 18 years

Inclusion criteria Module 6:

* The participant needs to be:

  1. a stakeholder within the community, state, region or country of the intervention who's position is related in any way to WASH in HCFs
  2. working in one of the intervention PHCFs. They do not need to be HCWs, they can also be hygiene technicians or in a leading position of the facilities.
* Minimum age of 18 years

Exclusion criteria:

Exclusion criteria Modules 1-3: HCW participants must not fulfil any of the following exclusion criteria:

* HCWs, whose primary occupation is not in the PHCF of the h4h project
* Suffering from any skin conditions not allowing the HCW to use soap or alcoholic hand rub
* Refusals to participate

Exclusion criteria Module 5: Refusals to participate.

Exclusion criteria Module 6: Refusals to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in handwashing practice with soap and water or hand sanitizer in the 5 critical moments of WHO | Up to 12 months
  The primary outcome is the number of times a participant performs good handwashing practice with soap or hand disinfectant at critical moments assessed by structured handwashing observations over an hour per unit in each health care facility. The number of critical moments serves as denominator. Critical moments are defined by the WHO as: i) Before touching a patient ii) Before clean/aseptic procedures iii) After risk/exposure to body fluids iv) After touching a patient v) After touching a patient's surroundings

SECONDARY OUTCOMES:
Change in self reported handwashing practice | Up to 12 months
  A) Self reported handwashing practice to answer for each critical moment on a five point Likert scale ranging from almost never to almost always with almost always being the better outcome.
Health care facilities: change in log-transformed number of total coliforms and E.coli | Up to 12 months
  B) The log-transformed number of total coliforms and E.coli CFUs per hand before handwashing
Experimental 1: Sum of incidences of absenteeism of work due to illness in health care workers | Up to 8 months
  C) The sum of incidences of absenteeism of work due to illness in health care workers per facility will be used as a measure for statistical analysis. The number of incidences will be measured with a diary approach: Every time this outcome takes place at facility level, it will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). The local study team is still discussing if a paper table, which will be collected once a month will be used as a diary, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.
Experimental 2: Sum of incidences of maternal mortality per health care facility | Up to 8 months
  D) The sum of incidences of maternal mortality per health care facility will be used as a measure for statistical analysis. The number of incidences will be measured with a diary approach: Every time this outcome takes place at facility level, it will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). The local study team is still discussing if a paper table, which will be collected once a month will be used as a diary, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.
Experimental 3: Sum of incidences of neonatal mortality per health care facility | Up to 8 months
  E) The sum of incidences of neonatal mortality per health care facility will be used as a measure for statistical analysis. The number of incidences will be measured with a diary approach: Every time this outcome takes place at facility level, it will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). The local study team is still discussing if a paper table, which will be collected once a month will be used as a diary, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.
Experimental 4: Sum of incidences of neonatal sepsis per health care facility | Up to 8 months
  F) The sum of incidences of neonatal sepsis per health care facility will be used as a measure for statistical analysis. The number of incidences will be measured with a diary approach: Every time this outcome takes place at facility level, it will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). The local study team is still discussing if a paper table, which will be collected once a month will be used as a diary, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.
Experimental 5: Sum of incidences of umbilical cord infections per health care facility | Up to 8 months
  G) The sum of incidences of umbilical cord infections per health care facility will be used as a measure for statistical analysis. The number of incidences will be measured with a diary approach: Every time this outcome takes place at facility level, it will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). The local study team is still discussing if a paper table, which will be collected once a month will be used as a diary, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.
Experimental 6: Sum of incidences of wound infection after stitching or surgical procedures per health care facility | Up to 8 months
  H) The sum of incidences of wound infection after stitching or surgical procedures per health care facility will be used as a measure for statistical analysis. The number of incidences will be measured with a diary approach: Every time this outcome takes place at facility level, it will be reported in a diary by the director of the PHCF (or someone who was appointed by the director). The local study team is still discussing if a paper table, which will be collected once a month will be used as a diary, or if alternatively, the team sends the doctor in charge once a month a mobile survey to fill in the data.

OTHER OUTCOMES:
Covariate 1: Age (age groups) | Up to 12 months
  The age groups are grouped into 18-24 years, 25-49 years and 50+ years and an option that the participant did not want to say to which group they belong.
Covariate 2: Education levels | Up to 12 months
  Education is measured in three levels according to the countries' education system: primary, secondary and superior education
Covariate 3: Sex | Up to 12 months
  Sex is measured in two groups: female and male. We did purposefully not ask about self-identified sex or gender with more than the two categories because in Mali and Burkina Faso this is an extremely sensitive issue which could lead to discrimination.
Covariate 4: Socio-economic status in income groups | Up to 12 months
  As it is not permitted to ask about income directly in the countries we work, we asked after the profession of the participant and their spouse and how many people live of their income. Our local partners will give us a rough estimate of the income which will be divided by the number of people living of it. We will test the model fit of this variable to see if it makes more sense to base it on two socio-economic status groups (low/high) or three groups (low/medium/high).
Covariate 5: Time since last training in hygiene (time groups) | Up to 12 months
  Time since last training in hygiene was assessed with the following time groups: 1-6 months ago, 6-12 months ago, more than 12 months ago and never had any training.
Covariate 6: Position in health care facility | Up to 12 months
  Job positions in the health care facilities were assessed according to common positions in the respective countries. Mali: medical doctor, public health nurse, obstetric nurse, midwife, intern, nursing assistant, matron, medical assistant, laboratory worker, vaccination agent, volunteers and other.
  Burkina Faso: medical doctor, nurse, midwife, patented birth attendant, auxiliary midwife, community health care workers, laboratory worker, intern, other.
Covariate 7: Water source of the health care facility | Up to 12 months
  The water source of the health care facility can be: no water source on premises, unprotected dug well, protected dug well, tubewell/borehole, piped supply outside the building, piped supply inside the building, other.

CONTACTS AND LOCATIONS:
Overall Officials: Mirko S. Winkler, Prof., Principal Investigator — Swiss Tropical and Public Health Institute and University of Basel
Locations (2):
- 24 community health centers (CSPS), Dédougou, Dédougou, Boromo, Burkina Faso
- 24 community health centers (CSCOMs), Ségou, Markala, Macina, Ségou, Tominian, Mali

IPD SHARING:
Plan to Share IPD: Yes
Coded or anonymized IPD can be shared internally with the following conditions:
  All rights, title and interest in and to research results shall be owned by the consortium member(s) whose personnel created such research results. Each consortium member has the right to use the research results of the other consortium member(s) for research purposes. Jointly generated research results are owned by the involved consortium members equally and can be used by all members. The use of data by third parties needs to be approved in writing by all consortium members.
  Once the project is officially terminated and the data has been published, all consortium members are free to conduct secondary data analysis provided there is no violation of ethical agreements and credits are properly acknowledged.
Supporting Information: Study Protocol
Time Frame: As our partner Terre des hommes actually collects the data in the field, they will have access to the IPD in real time in order to guaranty quality control. Other consortium members can receive the coded IPD if needed upon request as soon as the data is complete and cleaned.
Access Criteria: Internally:
  Data collected through ODK or KoboToolbox are stored on the ODK central server, to which the data collecting organization (Tdh, CESVI), RANAS and Swiss TPH have direct access. Other consortium members wishing to have access to data can directly contact someone with access to the server and ask them for the coded data.
  Externally:
  The use of data by third parties needs to be approved in writing by all consortium members.

REFERENCES:
- [Derived] Galli A, Ma'ani Abuzahra Y, Banziger C, Ballo A, Friedrich MND, Gross K, Harter M, Hattendorf J, Peter M, Tamas A, Owen BN, Winkler MS. Assessing the Effectiveness of a Multicomponent Intervention on Hand Hygiene and Well-Being in Primary Health Care Centers and Schools Lacking Functional Water Supply in Protracted Conflict Settings: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 3;13:e52959. doi: 10.2196/52959. PMID 38569182
- See also: Hands4health project website — https://hands4health.dev/
- See also: Gravit'eau Website — https://www.graviteau.ch/
- See also: RANAS Ltd. Website — https://www.ranasmosler.com/ranas
- See also: WASH FIT Website — https://washfit.org/#/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT05946980/Prot_SAP_000.pdf